CLINICAL TRIAL: NCT04314180
Title: Artificial Intelligence System for Assessing Image Quality of Slit-Lamp Images and Its Effects on Diagnosis: A Clinical Trial
Brief Title: Artificial Intelligence System for Assessing Image Quality of Slit-Lamp Images and Its Effects on Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Other Study IDs: IMAQUA2020-China-02
Record Dates: First submitted 2020-03-16; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Anterior Segment Disorders; Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Slit-lamp image quality assessment: Device: an artificial intelligence system for quality assessment of slit-lamp images. These patients are enrolled in primary healthcare units or the AI clinic at Zhongshan Ophthalmic Center
  Interventions: Device: Taking slit-lamp images

INTERVENTIONS:
Device: Taking slit-lamp images — The participant only needs to take several slit-lamp images as usual.

SUMMARY:
Slit-lamp images are widely used in ophthalmology for the detection of cataract, keratopathy and other anterior segment disorders. In real-world practice, the quality of slit-lamp images can be unacceptable, which can undermine diagnostic accuracy and efficiency. Here, the researchers established and validated an artificial intelligence system to achieve automatic quality assessment of slit-lamp images upon capture. This system can also provide guidance to photographers according to the reasons for low quality.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be aware of the contents and signed for the informed consent.

Exclusion Criteria:

* 1. Patients who cannot cooperate with a photographer such as some paralytics, the patients with dementia and severe psychopaths.
* 2. Patients who do not agree to sign informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion Criteria: - Patients should be aware of the contents and signed for the informed consent. Exclusion Criteria: - 1. Patients who cannot cooperate with a photographer such as some paralytics, the patients with dementia and severe psychopaths. - 2. Patients who do not agree to sign informed consent
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Performance of artificial intelligence system for distinguish between good image quality and poor image quality | 3 months
  Area under the receiver operating characteristic curves, sensitivity, specificity, positive and negative predictive values,accuracy

SECONDARY OUTCOMES:
The comparison of the performance for previous artificial intelligence diagnostic system with slit-lamp images of different image quality | 3 months
  Cohen's kappa coefficient, P value and other related statistic results

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No